CLINICAL TRIAL: NCT05794932
Title: Exercise Tolerance After Venous Recanalization for Post-thrombotic Syndrome: ETERecaVSPT
Brief Title: Exercise Tolerance After Venous Recanalization for Post-thrombotic Syndrome
Acronym: ETERecaVSPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0560
Record Dates: First submitted 2023-03-17; First posted 2023-04-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Post Thrombotic Syndrome; Venous Thromboses; Claudication, Intermittent
Keywords: iliac vein; inferior vena cava; exercice tolerance; cardio-pulmonary exercice testing; muscle physiological testing
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis; Intermittent Claudication | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stress test (Experimental): All patients will undergo a stress test before and after venous recanalization.
  Interventions: Diagnostic Test: Stress test

INTERVENTIONS:
Diagnostic Test: Stress test — Diagnostic Test:
  * Maximum effort test (CPET) on a cycloergometer
  * Leg muscle strength assessment
  * Leg muscle mass, composition and water compartments (segmental bioelectrical impedance)
  * Spirometry, arterial blood gaz, NO/CO transfer

SUMMARY:
Post-thrombotic syndrome (PTS) is the most frequently observed chronic complication of deep vein thrombosis (DVT), with an estimated cumulative incidence of 20-50%. Endovascular venous recanalization with angioplasty and stenting of obstructive lesions is the recommended treatment option to reduce or correct the symptoms of DVT. However, its impact on the physical capacity and breathlessness of patients has not been fully demonstrated. The heterogeneous evidences of clinical improvement is probably related to the presence or absence of collateral veins developed in these patients with proximal venous obstruction (iliac or iliofemoral with or without inferior vena cava involvement), which ensure the cardiac venous return. The aim of this study is to compare changes in maximal oxygen uptake after endovascular venous recanalization in DVT patients and to evaluate the hemodynamic, respiratory and muscular improvement induced by the restoration of venous flow in the occluded segments.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for endovascular treatment for post-thrombotic syndrome in a chronic context (6 months after the occurrence of thrombosis, without time limit), after validation of the indication during a monthly medical-radiological PCR (St Eloi vascular medicine team and vascular radiologist performing the endovascular treatment)
* Age >= 18 years

Exclusion Criteria:

* Contraindication to the performance of a maximal effort test on a cyclo-ergometer
* Refusal of consent after information
* Adult protected by law (guardianship, curatorship)
* Pregnant or breastfeeding woman
* Patient not affiliated to a social security system or not benefiting from such a system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
VO2 max | From baseline and 8 weeks
  Change in VO₂ max is the maximum (max) rate (V) of oxygen (O₂) the body is able to use during exercise from baseline to 8 weeks. It is measured in liters of O2 per minute

SECONDARY OUTCOMES:
Maximum aerobic power (in Watts) | From baseline and 8 weeks
  Maximum aerobic power is measured in watts before and after venous recanalization
Isowork power | From baseline and 8 weeks
  The isowork power is the power output assessed at the V'O2max before recanalization
Maximal exercise cardiac output (in litres per minute) | From baseline and 8 weeks
  Maximal exercise cardiac output is the cardiac output assessed by thoracic impedance et peak exercise before and after venous recanalization
Exercise change in Inspiratory capacity (in litres) | From baseline and 8 weeks
  Exercise change in Inspiratory capacity is the change between rest and peak exercise of the inspiratory capacity (the volume between end-expiratory volume and total lung capacity) before and after venous recanalization
Maximal exercise capillary volume (in millilitres) | From baseline and 8 weeks
  Maximal exercise capillary volume is the capillary volume at peak exercise assessed by NO/CO transfer before and after venous recanalization
Maximal exercise O2 arterial pressure (PaO2, in mmHg) | From baseline and 8 weeks
  Maximal exercise O2 arterial pressure is the oxygen partial pressure in the arterial blood, assessed at peak exercise, before and after venous recanalization
Maximal isometric torque during leg extension (in Newton.meters) | From baseline and 8 weeks
  Maximal isometric strength during leg extension is the maximal torque of the leg extension at 90° knee flexion assessed by a torque sensor before and after venous recanalization
Lower limb extracellular/total water (in %) | From baseline and 8 weeks
  Lower limb extracellular/total water is the water volume int the body compartments in each lower limb, assessed by a segmental bioelectrical impedancemeter before and after venous recanalization

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Arnaud de Villeneuve - CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No